CLINICAL TRIAL: NCT06622941
Title: A Multicenter, Open-label, Uncontrolled Phase II Study to Investigate Efficacy and Safety of ONO4538 in Patients With Rhabdoid Tumor
Brief Title: Study to ONO-4538 in Patients With Rhabdoid Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-126; jRCT2051240150 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Rhabdoid Tumor
MeSH Terms: conditions — Rhabdoid Tumor | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ONO-4538 (Experimental)
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538 — every 2 weeks
  Other Names: Nivolumab

SUMMARY:
Investigate the efficacy and safety of ONO-4538 for the treatment of rhabdoid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Not specified
2. Age (at the time of consent): 1 year or older
3. Patients who are refractory or intolerant to one or more regimens of chemotherapy for rhabdoid Tumors
4. Patients with advanced or recurrent rhabdoid Tumors not eligible for curative resection

Exclusion Criteria:

1. Patients with a history of active concurrent malignancy or complications
2. Patients with spinal lesions expected to require radiation therapy or surgical intervention during the trial period
3. Patients with concomitant central nervous system disorders other than AT/RT that are inadequately controlled or may lead to discontinuation of the investigational drug

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 4.5 years

SECONDARY OUTCOMES:
Objective response rate (ORR) (site investigator assesment) | up to 4.5 years
Overall survival (OS) | up to 4.5 years
Progression free survival (PFS) | up to 4.5 years
Disease control rate (DCR) | up to 4.5 years
Time to response (TTR) | up to 4.5 years
Best overall response (BOR) | up to 4.5 years
Percent change from baseline in the sum of diameters of target lesions | up to 4.5 years
Best reduction percent change from baseline in the sum of diameters of target lesions | up to 4.5 years
Incidence of Adverse Events [Safety] | Up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (4):
- Japan (4):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Osaka City General Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No